CLINICAL TRIAL: NCT03624933
Title: Effects of Extended Cannabis Abstinence on Symptoms and Cognition in Depressed Individuals
Brief Title: Effects of Cannabis Abstinence on Symptoms and Cognition in Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Tony George, Chief, Addictions Division, Centre for Addiction and Mental Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 069/2017
Record Dates: First submitted 2018-07-25; First posted 2018-08-10 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-09

CONDITIONS: Cannabis Use Disorder; Major Depressive Disorder; Cognition
Keywords: Depression; Cognitive Functioning; Cannabis Use Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Intervention Model Description: This is an open label intervention of contingent reinforcement and behavioral support to try to enhance cannabis abstinence for 28 days with people with Major Depressive Disorder. We will analyze data post hoc from this study as a function of subjects who attain abstinence versus those who do not.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 28-Day Cannabis Abstinence (Experimental): The study will assess the changes that occur after a 28-day abstinence period in patients with Major Depressive Disorder (MDD) and comorbid Cannabis Use Disorder (CUD). Patients will be instructed to initiate abstinence 12 hours prior to the baseline session and will come in for weekly visits involving a series of clinical, cognitive, and substance use assessments.
  Interventions: Behavioral: Weekly Behavioral Coaching Session; Behavioral: Contingency Management

INTERVENTIONS:
Behavioral: Weekly Behavioral Coaching Session — The participants will be provided with a 20-minute individual behavioral support session weekly for 4 weeks (28 days of abstinence), designed to provide them with tools and techniques to manage the craving and withdrawal symptoms that occur with cessation.
Behavioral: Contingency Management — If the participant's weekly abstinence is successful as determined by the urine results on day 28, the participant will receive an additional $300.00 cash bonus on top of their hourly $10 compensation for attending all visits. We predict that this cash bonus is enough incentive to allow for the behavioural change of abstinence in this patient population.

SUMMARY:
The objective of this study is to assess the changes in symptoms and cognition that occur after a 28-day abstinence period in patients with comorbid Cannabis Use Disorder (CUD) and Major Depression (MDD). This study employs a 28-day abstinence paradigm a total of 8 visits to the CAMH Russell site (screening, training, baseline, week 1, week 2, week 3, week 4, follow-up). Participants should be between the ages of 18-55, meet criteria for moderate depression and CUD, be non-treatment seeking, and be on a stable dose of antidepressant medication. The study visits will take up a total of approximately 22.5 hours with compensation for time provided. These visits will involve multiple clinical, substance use, and cognitive assessments. Abstinence will be maintained by weekly behavioural coaching sessions and contingency reinforcement.

ELIGIBILITY:
Inclusion Criteria:

* ages 18-55
* meet DSM-5 diagnostic criteria for cannabis use disorder (cannabis use >1 g/day, CUDIT score >12)
* meet DSM-5 diagnostic criteria for Major Depressive Disorder as determined using the SCID
* be an outpatient receiving a stable dose of antidepressant medication(s) for at least 1 month
* have a Hamilton Depression Rating Scale (HDRS-17) baseline total score greater than 14
* have a Full Scale IQ greater than 80 as determined by the WTAR
* be a non-treatment seeking cannabis user
* evidence of sufficient motivation and effort as measure by a Test of Memory Malingering (TOMM) score greater than 45
* urinary baseline THC-COOH levels greater than 150 ng/ml

Exclusion Criteria:

* meets criteria for abuse or dependence of alcohol or other illicit substances within the part 6 months (with the exception of cannabis, nicotine, or caffeine)
* positive urine screen for illicit substances other than cannabis, nicotine or caffeine
* current suicidal or homicidal ideation
* psychotic disorder diagnosis (e.g. schizoaffective disorder, major depression with psychotic features) as determined by the SCID
* head injury with loss of consciousness greater than 2 minutes or requiring hospitalization
* neurological or medical condition determined to effect cognition
* be treatment seeking for cannabis use

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
The effects of 28 day cannabis abstinence on change in depressive symptoms in cannabis-dependent patients with Major Depressive Disorder (MDD) as assessed by the Hamilton Rating Scale for Depression (HRSD). | Weekly (Day 0, Day 7, Day 14, Day 21, Day 28) and at 8 weeks (Follow-up Day 56)
  The clinical assessment will be administered weekly during the abstinence period and conducted by study personnel. The HRDS is used to evaluate depression on a 17-item scale with higher values indicating worse depressive symptoms.

SECONDARY OUTCOMES:
The effects of 28 day cannabis abstinence on change in cognitive function in cannabis dependent patients with Major Depressive Disorder (MDD) as assessed by a cognitive battery administered at Baseline, Week 2, Endpoint and Follow-Up. | Bi-Weekly (Day 0, Day 14, Day 28) and at 8 Weeks (Follow-up Day 56)
  The cognitive battery will include the primary outcome of verbal memory (assessed by Hopkins Verbal Learning Test) and will be compared to baseline (Day 1) performance. Cortical inhibition will also be assessed and compared.
The effects of 28 day cannabis abstinence on change in co-occurring anxiety in cannabis dependent patients with MDD as assessed by the Beck Anxiety Inventory (BAI) administered weekly. | Weekly (Day 0, Day 7, Day 14, Day 21, Day 28) and at 8 weeks (Follow-up Day 56)
  The clinical assessment will be administered at Baseline, weekly during the abstinence period and Follow-up and will be conducted by study personnel. The BAI is a 21-item scale used to evaluate the severity of anxiety symptoms with higher values indicating worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Tony George, M.D., FRCPC, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Sorkhou M, Rabin RA, Rabin JS, Kloiber S, McIntyre RS, George TP. Effects of 28 days of cannabis abstinence on cognition in major depressive disorder: A pilot study. Am J Addict. 2022 Sep;31(5):454-462. doi: 10.1111/ajad.13305. Epub 2022 Jun 11. PMID 35690891